CLINICAL TRIAL: NCT02993575
Title: Pharmacokinetics of Flucloxacillin Given by Continuous or Intermittent Infusion as Therapy to Patients With an Infection in the Intensive Care Unit (ICU)
Brief Title: Pharmacokinetics of Flucloxacillin Given by Continuous or Intermittent Infusion to ICU Patients
Acronym: FANATIC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Rijnstate Hospital (Other); UMC Utrecht (Other); Tergooi Hospital (Other); Gelderse Vallei Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF-16.08
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Bacterial Infections
Keywords: Pharmacokinetics; Flucloxacillin; Continuous infusion; Intensive Care Unit
MeSH Terms: conditions — Bacterial Infections | interventions — Floxacillin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for determination of total flucloxacillin and free flucloxacillin
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Flucloxacillin — Dose according to summary of product characteristics (SPC) or local protocols: intermittent and continuous infusion
  Other Names: Floxapen

SUMMARY:
The pharmacokinetics of flucloxacillin are expected to be different in ICU patients compared to non-ICU patients. The investigators will determine total and free flucloxacillin concentrations in 30 ICU patients, who will get continuous (n=10) or intermittent infusion (n=20) of flucloxacillin as standard care.

Full pharmacokinetic curves will be taken for individual patients on the intermittent dosing regimen and limited sampling will be taken for individual patients on the continuous dosing regimen on day 2 and 4.

DETAILED DESCRIPTION:
The pharmacokinetics of flucloxacillin are expected to be different in ICU patients compared to non-ICU patients. There is a substantial risk that present standard dosing regimens of antibiotics lead to suboptimal outcomes for patients on the ICU. To prevent the risk of inadequate dosing in critically ill patients, it is important to optimize dosing regimens in ICU patients.

With this study the investigators will define pharmacokinetics of flucloxacillin in ICU patients and search for variables influencing pharmacokinetics. By using population modeling the investigators will simulate different dosing regimens, intermittent and continuous, and compare probability of target attainment between continuous and intermittent infusion.

To be able to include 30 patients within the study duration, a multi-centre approach is necessary.

Patients will receive standard care, as stated in the product characteristics or according to local protocols. Minimally invasive blood sampling for pharmacokinetic analysis will be retrieved through a central venous catheter or an arterial line. Full pharmacokinetic curves will be taken for individual patients on the intermittent dosing regimen and limited sampling will be taken for individual patients on the continuous dosing regimen on day 2 and 4.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to an ICU
2. Subject is at least 18 years old on the day of the first dosing
3. Is managed with a central venous catheter or arterial line
4. Patient is treated with flucloxacillin

Exclusion Criteria:

1. Has previously participated in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving flucloxacillin for treating a suspected or proven bacterial infection at the ICU will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Clearance | Day 2 and 4
  Full pharmacokinetic curves will be taken on Day 2 and Day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No